CLINICAL TRIAL: NCT02825784
Title: A Multicenter, Open Label, Uncontrolled Study to Evaluate the Acceptability, Tolerability and Nutritional Suitability of Renastart: Specially Formulated to Meet the Unique Nutritional Needs From Birth to 10 Years With Chronic Kidney Disease
Brief Title: A Multicenter Study to Evaluate the Nutritional Suitability of Renastart
Acronym: Renastart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA-REN-072013-03
Record Dates: First submitted 2016-06-17; First posted 2016-07-07 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Disease; Hyperkalemia
Keywords: potassium chronic kidney disease CKD children
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renastart (Experimental): Compared to cows' milk and/or standard pediatric enteral feeds, Renastart has the following additional nutritional features that are beneficial in children with CKD: lower phosphorus, calcium and vitamin A. The powder presentation allows flexibility with dilutions to facilitate the provision of adequate energy and protein to support growth in children with CKD.
  For each subject, the recommended daily intake of Renastart is determined by the dietitian in collaboration with the local PI and primary nephrologist based on individual nutritional requirements, specifically dietary intake of potassium and serum potassium levels.
  Renastart is to be given by the clinician and based on clinical and nutritional needs. Standard preparation guidelines can be found on the Renastart label.
  Interventions: Dietary Supplement: Renastart

INTERVENTIONS:
Dietary Supplement: Renastart — Renastart: specially formulated to meet the unique nutritional needs of children from birth to 10 years with chronic kidney disease (CKD).

SUMMARY:
A multicenter, open label, uncontrolled study to evaluate the acceptability, tolerability, and nutritional suitability of a medical food (Renastart, Vitaflo International Ltd) specially formulated to meet the unique nutritional needs of children from birth to 10 years with chronic kidney disease (CKD)

DETAILED DESCRIPTION:
A multicenter, open label, uncontrolled study to evaluate the acceptability, tolerability, and nutritional suitability of a medical food (Renastart, Vitaflo International Ltd) specially formulated to meet the unique nutritional needs of children from birth to 10 years with chronic kidney disease (CKD)

Primary Objective To investigate the nutritional suitability of Renastart in children aged 10 years and under with CKD, particularly with respect to the dietary management of hyperkalemia and the maintenance / improvement of growth.

Secondary Objectives To investigate the acceptance, compliance, palatability, and tolerance of Renastart in children aged under 10 years with CKD.

A total of 15 children with CKD will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 10 years or under at the time of enrolment into the study.
2. Diagnosed with Chronic Kidney Disease
3. Requirement for a low potassium diet, as evidence by elevated serum potassium levels (> normal reference value which is 3.5-5.0 mmol/L)
4. Requirement for a low potassium enteral formula to provide a minimum of 20% of daily energy (kcal) requirements. (calculated according to individual child's needs and according to local clinical practice)
5. Written informed consent provided by parent/primary caregiver.
6. Assent provided by child, if appropriate.

Exclusion Criteria:

1. Receiving total parenteral nutrition (TPN).
2. Intolerance or allergy to cow's milk or any other ingredients in Renastart.
3. Prior intolerance of Renastart formula.
4. Any disorders which in the investigator's opinion may cause significant gastrointestinal malabsorption.
5. Liver failure.
6. Active infection or presenting with any signs or symptoms of an infectious disease at screening.
7. Concurrent enrollment into another clinical trial.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in serum potassium level | Baseline, week 8, week 16
  To evaluate the nutritional suitability of Renastart, specifically in relation to management of hyperkalemia via blood tests

SECONDARY OUTCOMES:
Change in height (cm) | Baseline, week 8, week 16
  To monitor the maintenance / improvement of growth over the course of the study.
Change in mass (kg) | Baseline, week 8, week 16
  To monitor the maintenance / improvement of growth over the course of the study.
Palatability | Throughout the 16 weeks
  To evaluate the palatability of Renastart when taken orally via a patient questionnaire.
Gastrointestinal tolerance | Throughout the 16 weeks
  To evaluate the GI tolerance of Renastart when taken orally or by enteral feeding tube via a patient questionnaire.
Compliance | Throughout the 16 weeks
  To evaluate patient compliance with Renastart administration when taken orally or by enteral feeding tube via a patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hoppe, Principal Investigator — Universitätsklinik Bonn
Locations (3):
- Germany (3):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Koln, Cologne
  - Universitatsklinikum Essen, Essen

IPD SHARING:
Plan to Share IPD: No